## The Effect of Intravenous Acetaminophen on Post-Operative Pain After Craniotomy (NCT03445390)

May 29, 2013

Mark Burbridge, MD, Principal Investigator Stanford University Stanford, California 94305

## Acetaminophen efficacy study protocol

## **Brief protocol:**

Patients will be consented for the study on the day of their first surgery.

Randomization will be coordinated with pharmacy. Patient will be randomized by pharmacy to receive either acetaminophen or placebo at the end of the case, and then for the next 24 hours.

Anesthesia will be induced with fentanyl, propofol, and rocuronium, administered at the discretion of the anesthesiologists.

The anesthetic will be maintained with a combination of isoflurane, remifentanil, nitrous oxide, and/or propofol.

The surgeons are free to infiltrate the incision with local anesthetic.

At the end of the case while the patient is emerging from anesthesia, administer 1 gram IV acetaminophen or placebo over 15 minutes. Except for remifentanil, do not administer any other opioids at the end of the case.

At arrival to the ICU, a patient controlled analgesia (PCA) pump will be setup and immediately made available to the patient.

The ICU nurse will be informed of the study, and handed material that will explain their portion of the study, including assessments and drug administration.

After 24 hours, the post-operative assessment form filled out by nursing will be collected.

Within 30 days of discharge following the second surgery, the patients will be contacted via their method of choice to participate in a brief survey.